CLINICAL TRIAL: NCT04774263
Title: The Acceptability of a Real-time Localization of Patients and Caregivers
Brief Title: The Acceptability of a Real-time Localization for Patients and Caregivers
Acronym: RTLS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Gerontopole Auvergne Rhone-Alpes (AURA) (Other); Saint Etienne School of Mine (Other)
Responsible Party: Sponsor
Other Study IDs: GA-2021-03
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Disease
Keywords: Acceptability study; new technologies; health sector; real time location system
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: general population
  Interventions: Other: Individual interviews
- emergency caregivers: emergency caregivers
  Interventions: Other: Individual interviews

INTERVENTIONS:
Other: Individual interviews — Discussion between the searcher and the participant about representations and acceptability about a potential real time localization system

SUMMARY:
Technological innovations are taking over our daily lives, particularly in the health sector. Real-time location systems for healthcare professionals and patients are developing in hospitals. Today few studies have focused on the acceptability of this new technology. The present research, which aims to study the acceptability of a real-time localization systems, reveals a definite utility and acceptability from the patient's point of view, subject to conditions. Indeed, the guarantee of data security and the concrete interest for the patient must be explained. For healthcare professionals working in emergency departments, the usefulness of new technologies in their work is now well established. Nevertheless, the acceptability of a real-time location systems received lukewarm reviews. It depends mainly on reticence linked to the fear of a possible deviation in the use of the data collected.

DETAILED DESCRIPTION:
study the acceptability of a real-time localization of patients and caregivers

ELIGIBILITY:
Inclusion Criteria:

* For general population : people have been hospitalized at least once
* For caregivers : works in emergency service

Exclusion Criteria:

* Person with a neurological disease
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population who have been hospitalized at least once and caregivers who works in emergency service
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
opinion and representations about a real time localization system | Days:30
  Measure by individual interviews

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Augusto, Study Director — augusto@emse.fr
Locations (1):
- Gérontopole AURA, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No